CLINICAL TRIAL: NCT02925676
Title: Evaluation of the Hypoglycaemia Notification Device Hyposafe H02 - the Pilot 2 Study - in Subjects With Type 1 Diabetes
Brief Title: Evaluation of the Hypoglycaemia Notification Device Hyposafe H02
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow recruitment
Sponsor: UNEEG Medical A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pilot 2 Diabetes
Record Dates: First submitted 2016-09-19; First posted 2016-10-06 (Estimated); Results first posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Hypoglycaemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- hyposafe H02 (Experimental): All subjects included are assigned to hyposafe H02-testing
  Interventions: Device: hyposafe H02

INTERVENTIONS:
Device: hyposafe H02 — hypoglycaemia notification device

SUMMARY:
To evaluate the technical performance of the hyposafe H02 during everyday activities and during insulin-induced hypoglycaemia, in addition to safety issues associated with the implantation and use of the hyposafe H02 in subjects with type 1 diabetes.

DETAILED DESCRIPTION:
While a finger prick test accurately measures the blood glucose level, it does not provide continuous measurements and hence it is unreliable as a hypoglycaemia notification. Recent studies have indicated that the use of continuous glucose monitoring (CGM) reduces the risk of severe hypoglycaemia. However, some find these devices troublesome to use and are annoyed by the inaccuracy of the measurements and even after short-term use the coverage in subgroups of patients is as low as 50% of the time. Thus, there is a medical need for a reliable hypoglycaemia notification which is easy and convenient to use and with high sensitivity and high rate of positive prediction.

This clinical investigation is designed to evaluate the sensitivity and the positive predictive value of the Hyposafe H02 in subjects with type 1 diabetes during everyday activities and during insulin-induced hypoglycaemia. In addition, the investigation provides information regarding safety and usability of the device. This to verify that the Hyposafe H02 works as intended in subjects with type 1 diabetes before proceeding with a larger study in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study related activities
* Type 1 diabetes diagnosed at least five years prior to inclusion in the study
* Impaired awareness and/or history of at least one severe hypoglycaemia within the preceding year

Exclusion Criteria:

* Severe cardiac disease
* History of stroke or cerebral haemorrhage and any other structural cerebral disease
* Active cancer or cancer diagnosis within the past 5 years
* Uraemia defined as s-creatinine ≥ 3 times upper reference value
* Liver disease defined as s-ALAT ≥ 3 times upper reference interval
* Epilepsy
* Use of antiepileptic drugs for any indication
* Clinically important hearing impairment
* Use of active implantable medical device including pacemaker and ICD-unit and cochlear implant
* Use of following drugs: Chemotherapeutic drugs of any kind, Methotrexate, Third generation antipsychotic drugs (aripiprazole, quetiapine, clozapine, ziprasidone, paliperidone, risperidone, sertindole, amisulpride, olanzapine)
* Contraindications to the local anaesthetic used during implantation
* Known or suspected abuse of alcohol or any other neuro-active substances
* Infection at the site of device implantation
* Any haemorrhagic disease
* Females of childbearing potential who are pregnant or intend to become pregnant or are not using adequate contraceptive methods throughout the study
* Performing extreme sport, including scuba diving (snorkel diving is allowed) or parachute jumping
* Incapable of understanding the subject information or unlikely to complete the study for any reason
* Operating MRI scanners
* Operating handheld transceivers for communication (e.g. within the police, medical, fire, air traffic control, marine or military)
* Working at broadcast stations for television or FM/DAB radio
* Use of CGM or FGM with visible glucose measurements and activated glucose notifications
* Involved in therapies with medical devices that deliver electrical energy into the area around the implant

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Pedersen-Bjergaard, MD, PhD, Principal Investigator — Nordsjaellands Hospital
Locations (2):
- Denmark (2):
  - North Zealand Hospital, Hillerød
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hyposafe H02
Started | 8
Completed | 7
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Hyposafe H02: All subjects included are assigned to hyposafe H02-testing
  hyposafe H02: hypoglycaemia notification device
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 8
Region of Enrollment [Number; unit: participants]
  Denmark | 8
Dieabetes duration [Mean (Standard Deviation); unit: years] | 35 (16.1)

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity
Description: Number of spontaneous hypoglycaemic episodes detected by the hyposafe H02 compared to the total number of validated spontaneous hypoglycaemic episodes. Validation was performed by self-measured blood glucose (SMBG).
Time Frame: 3 months
Measure: Number; unit: Percentage
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Percentage
  Sensitivity (day) | 100
  Sensitivity (night) | 100

2. Primary Outcome: Positive Predictive Value
Description: Number of validated spontaneous hypoglycaemic episodes detected by the hyposafe H02 compared to the total number of notification from the hyposafe H02. Validation was performed by self-measured blood glucose (SMBG).
Time Frame: 3 months
Measure: Number; unit: Percentage
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Percentage
  Positive predictive value (day) | 8
  Positive predictive value (night) | 2

3. Secondary Outcome: Overall Sensitivity
Description: Total number of hypoglycaemic episodes detected by the hyposafe H02 compared to the total number of validated hypoglycaemic episodes. Validation was performed by self-measured blood glucose (SMBG) or plasma glucose (PG).
Time Frame: 3 months
Measure: Number; unit: Percentage
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Percentage | 81

4. Secondary Outcome: Overall Positive Predictive Value
Description: Total number of validated hypoglycaemic episodes detected by the hyposafe H02 compared to the total number of alerts from the hyposafe H02. Validation was performed by self-measured blood glucose (SMBG) or plasma glucose (PG).
Time Frame: 3 months
Measure: Number; unit: Percentage
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Percentage | 11

5. Secondary Outcome: Sensitivity During Insulin-induced Hypoglycaemia
Description: Number of insulin-induced hypoglycaemic episodes detected by the hyposafe H02 compared to the total number of insulin-induced hypoglycaemic episodes.
Time Frame: 2 days
Measure: Number; unit: Percentage
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Percentage | 57

6. Secondary Outcome: Positive Predictive Value for Insulin-induced Hypoglycaemia
Description: Number of insulin-induced hypoglycaemic episodes detected by the hyposafe H02 compared to the total number of alerts from the hyposafe H02
Time Frame: 2 days
Measure: Number; unit: Percentage
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Percentage | 100

7. Secondary Outcome: Number of Participants With a Satisfactory EEG Quality Test
Description: The EEG quality test was performed twice in the study. At start up and at the end of the study. Evaluation was based on visual review of EEG of known phenomena and artefacts by an experienced EEG reviewer.
Time Frame: start up and after 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Participants | 7

8. Secondary Outcome: Change in Impedance (kOhm) Over Time
Description: The EEG performance was measured as the impedance as a function of time. An impedance value below 5 kOhm is considered very good. Number of participants with impedance values below 5 kOhm and no change over time is reported.
Time Frame: start up and after 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Participants | 7

9. Secondary Outcome: Device Deficiencies
Description: Total number of device deficiencies
Time Frame: 4 months
Measure: Number; unit: Counts
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 8
Counts | 15

10. Secondary Outcome: Mean Glucose Level at the Time of a Hypoglycaemia Notification
Description: Glucose levels were measured at the time of a hypoglycaemia notification during an outpatients settings (the spontaneous episodes) and during insulin-induced hypoglycaemia (the insulin-induced episodes)
Time Frame: 3 months
Measure: Mean (Full Range); unit: mmol/L glucose
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
mmol/L glucose
  Spontanous episodes | 2.4 [1.9 to 3.8]
  Insulin-induced episodes | 2 [1.7 to 2.6]

11. Secondary Outcome: Development in Discomfort Over Time Based on Questionnaires
Description: Implant discomfort over time were evaluated at 3 time points; on average 3 weeks, 7 weeks and 15 weeks after implantation (baseline). Here the categories were converted into cardinal numbers: ranging from strongly agree=5 to strongly disagree=1 on the statement ''The implant has not caused discomfort in the past two days'.
Time Frame: 3 weeks, 7 weeks and 15 weeks after implantation (baseline)
Measure: Mean (Full Range); unit: Score on a scale
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Score on a scale
  3 weeks after implantation | 4.1 [3 to 5]
  7 weeks after implantation | 4.7 [4 to 5]
  15 weeks after implantation | 4.9 [4 to 5]

12. Secondary Outcome: User Satisfaction Based on Questionnaire
Description: User satisfaction were evaluated as to whether the subjects wished to continue to use the device
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Participants
  Number of participants that would like to continue to use the device | 2
  Number of participants that would not like to continue to use the device | 5

13. Secondary Outcome: Mean Number of Hours of Use Per Device
Description: Mean number of hours of use per device is measured as recording time of device
Time Frame: 3 months
Measure: Mean (Full Range); unit: Hours
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Hours
  Use per day | 13.5 [11.5 to 15.9]
  Use per night | 8.2 [6.8 to 11]

14. Secondary Outcome: Response to Hypoglycaemia Notification
Description: Response to hypoglyceamia notifications measured as the participants were able to take preventive actions upon notification of hypoglycaemia in an outpatient settings (the spontaneous hypoglycemic episodes) and during insulin-induced hypoglycaemia
Time Frame: 3 months
Measure: Number; unit: Percentage
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 7
Percentage
  Spontaneous hypoglycemic episodes | 100
  Insulin-induced hypoglycemic episodes | 87.5

15. Secondary Outcome: Alarm Fatigue Based on Questionnaire
Description: The participants were given a questionnaire regarding their preferences for sensitivity and false alarms at the end of the study. Reporting are for preferences during the day.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Overall Study: Hyposafe H02
Number analyzed (Participants) | 5
Participants
  95% sensitivity - 15 false notifications weekly | 2
  90% sensitivity - 9 false notifications weekly | 3

ADVERSE EVENTS:
Time Frame: Adverse event were collected in a period of 17 weeks for each participant
Description: The adverse events were defined according to ISO14155:2011
Arm/Group | Overall Study: Hyposafe H02
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 8/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Overall Study: Hyposafe H02 (N=8)
Skin infection (Skin and subcutaneous tissue disorders) | 1 (2) — Possible or probable related to device
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) — Possible or probable related to device
Implant site pain (General disorders) | 5 (8) — Administration site conditions Possible or probable related to device
Ear pain (Ear and labyrinth disorders) | 1 (1) — Possible or probable related to device
Implant site hyperesthesia (Nervous system disorders) | 1 (1) — Possible or probable related to device
Hypoglycaemia (Endocrine disorders) | 1 (1) — Possible or probable related to device
Thooth infection (Infections and infestations) | 1 (3) — Unlikely related to device
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 (1) — Unlikely related to device
Urinary tract infection (Infections and infestations) | 1 (2) — Unlikely related to device
Influenza (Infections and infestations) | 1 (1) — Unlikely related to device
Renal stone removal (Surgical and medical procedures) | 1 (1) — Unlikely related to device

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review. The sponsor extend the embargo with up to 90 days if filling a patent is wanted by the Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-16): https://cdn.clinicaltrials.gov/large-docs/76/NCT02925676/Prot_SAP_000.pdf